CLINICAL TRIAL: NCT06667141
Title: ACR-2316-101: Phase 1 Study of ACR-2316 in Subjects With Advanced Solid Tumors
Brief Title: Phase 1 Study of ACR-2316 in Specific Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Acrivon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACR-2316-101
Record Dates: First submitted 2024-10-23; First posted 2024-10-31 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Specific Advanced Solid Tumors
Keywords: ACR-2316; WEE1; PKMYT1; Locally advanced, recurrent or metastatic solid tumors; P53
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies; Recurrence

STUDY DESIGN:
Intervention Model Description: Dose escalation - Evaluable participants for dose limiting toxicity (DLT), maximum tolerated dose (MTD) determination for ACR-2316 administered per cohort
  Dose expansion - participants with certain tumor types will be randomized 1:1 to receive1 of the 2 dose levels that will be selected for the determination of RP2D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): ACR-2316 will be administered using a 3-week or a 4-week schedule.
  Interventions: Drug: ACR-2316
- Dose expansion (Experimental): ACR-2316 will be administered using a 3-week or a 4-week schedule.
  Interventions: Drug: ACR-2316

INTERVENTIONS:
Drug: ACR-2316 — ACR-2316 is an experimental drug

SUMMARY:
This is a first in-human, Open-label Phase 1 study to assess the safety of ACR-2316 for the treatment of subjects with specific, histologically confirmed, locally advanced, recurrent or metastatic solid tumors.

DETAILED DESCRIPTION:
The Phase 1 monotherapy clinical trial for ACR-2316 is designed to assess the safety and tolerability of ACR-2316. Additional objectives include the determination of the maximal tolerated dose and recommended Phase 2 monotherapy dose, characterization of the pharmacokinetic profile and pharmacogenomics, and preliminary evaluation of anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Histologically or cytologically proven metastatic, recurrent or locally advanced selected solid tumors.
3. Must be willing to provide redacted pathology report.
4. Subjects should have received no more than 3 lines of systemic therapy for recurrent disease.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at trial entry and an estimated life expectancy of at least 3 months.
6. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST v1.1.
7. Adequate organ functions.
8. Must have progressed after prior line of treatment.

Exclusion Criteria (all participants):

1. Participants with known symptomatic brain metastases.
2. Participant had systemic therapy within 3 weeks prior to the first dose of study drug.
3. Participant had radiation therapy for curative intent within 4 weeks prior to the first dose of study drug.
4. Participant had palliative radiation therapy within 2 weeks prior to the first dose of study drug.
5. Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-08-12 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation | Number of DLT events during the DLT observation period (up to 28 days)
  To determine the MTD of ACR-2316.
Dose Expansion | RP2D supported by safety, PK, PD, and emerging clinical activity data through study completion, an average of 1 year.
  To determine the RP2D of ACR-2316.
Dose Expansion | Incidence and grades of TEAEs and TRAEs per NCI CTCAE v.5.0 and number of dose decreases, number of dose delays, and SAEs through study completion, an average of 1 year.
  To assess the safety and tolerability of ACR-2316
Dose Expansion | Confirmed ORR per Recist v1.1 and DOR, CBR, assessed every 6 weeks from baseline thorough study completion, an average 1 year or until death.
  To determine preliminary anti-tumor activity of ACR-2316.

SECONDARY OUTCOMES:
Dose Escalation | This will be evaluated through study completion, an average of 1 year.
  To assess the safety and tolerability of ACR-2316. Safety will be assessed by the incidence of AEs characterized overall and by type, incidence, severity graded according to NCI CTCAE v5.0, seriousness, and relationship to study treatment.
Dose Escalation | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: maximum plasma drug concentration (Cmax).
Dose Escalation | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: minimum plasma drug concentration (Cmin).
Dose Escalation | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: time to maximum plasma drug concentration (tmax).
Dose Escalation | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: time of last quantifiable plasma drug concentration (tlast).
Dose Escalation | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: area under the plasma concentration versus time curve (AUC).
Dose Escalation | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: plasma drug concentration at 24 hours post-dose (C24).
Dose Escalation | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: apparent volume of distribution (Vz/F).
Dose Escalation | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: terminal elimination half-life (t½).
Dose Escalation | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: apparent oral clearance (CL/F).
Dose Expansion | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: maximum plasma drug concentration (Cmax).
Dose Expansion | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: minimum plasma drug concentration (Cmin).
Dose Expansion | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: time to maximum plasma drug concentration (tmax).
Dose Expansion | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: time of last quantifiable plasma drug concentration (tlast).
Dose Expansion | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: area under the plasma concentration versus time curve (AUC).
Dose Expansion | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: plasma drug concentration at 24 hours post-dose (C24).
Dose Expansion | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: apparent volume of distribution (Vz/F).
Dose Expansion | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: terminal elimination half-life (t½).
Dose Expansion | Pharmacokinetic (PK) testing in Cycle 1, 2 & 3 (each cycle is up to 28 days). Predose and multiple time points after dose up to Cycle 3.
  To assess Pharmacokinetics: apparent oral clearance (CL/F).

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - HonorHealth Research Institute, Phoenix, Arizona
  - Precision NextGen Oncology & Research Center, Beverly Hills, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Denver Health One, Denver, Colorado
  - Florida Cancer Specialist, Sarasota, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Montefiore Medical Centre, The Bronx, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - Tennessee Oncology, Franklin, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - Next Virginia, Fairfax, Virginia